CLINICAL TRIAL: NCT06607536
Title: Clinical Effectiveness of the Calcium Chloride (CaCl2) Surface- Treated Orthodontic Mini Implant (OMI) in a Split-Mouth Randomised Controlled Trial (RCT)
Brief Title: Clinical Effectiveness of the Calcium Chloride (CaCl2) Surface- Treated Orthodontic Mini Implant (OMI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Suzanne Husun Reginald Iggan, Dr, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/09/2021 (FB/56)
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Basic Science; Orthodontic Appliance Complication; Malocclusion
Keywords: orthodontic mini implant; surface treated; anchorage; orthodontics
MeSH Terms: conditions — Malocclusion | interventions — Denture, Partial, Fixed, Resin-Bonded

STUDY DESIGN:
Intervention Model Description: 3 arm parallel, split mouth
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: sealed envelop
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Calcium Chloride (Experimental): Mini implant immersed in the calcium chloride 0.1M solution
  Interventions: Other: calcium chloride surface treatment in mini implant
- Acid Etch (Active Comparator): mini implant etched with hydrochloric acid
  Interventions: Other: Acid Etched
- machined mini implant (No Intervention): non surface treated mini implant

INTERVENTIONS:
Other: calcium chloride surface treatment in mini implant — 0.1M of Calcium Chloride were used to immersed the orthodontic mini implant
  Arms: Calcium Chloride
Other: Acid Etched — Mini implant etched in Hydrochloric acid
  Arms: Acid Etch

SUMMARY:
The goal of this split mouth, randomised control study was to compare the clinical effectiveness of surface treated Calcium Chloride orthodontic mini implant in orthodontic patients. The main question[s] it aimed to answer were:

Does the clinical effectiveness based on overall stability in maximum insertion torque and maximum removal torque measurement vary between untreated surface OMI, treated surface OMI with acid etching only and treated surface OMI with acid etching and calcium chloride immersion?, Does the surface roughness of OMI surface post removal vary between untreated surface OMI, treated surface OMI with acid etching only and treated-surface MI with acid etching and calcium chloride immersion? Does the success rate vary between untreated surface OMI, treated surface OMI with acid etching only and treated surface OMI with acid etching and calcium chloride immersion?Does the oral health quality of life and pain vary between untreated surface OMI, treated surface OMI with acid etching only and treated surface OMI with acid etching and calcium chloride immersion? Participants who is eligible for the study , orthodontic patient requiring moderate to high anchorage will be allocated to 2 groups (Group 1 : calcium chloride and control, Group 2 : acid etch, and control) to be used during the orthodontic treatment. The intervention is calcium chloride; the Calcium Chloride, positive control is the acid-etched and control is the machined group OMI. Comparison of the maximum insertion and removal torque, oral health quality of life, success rate and the surface roughness between the different groups of OMI.

DETAILED DESCRIPTION:
1.1 Study Design A triple-blinded, three-arm parallel-group randomized controlled trial was conducted at a single center. The trial assesses the effectiveness of an intervention through a split-mouth clinical study design.

1.2 Study Duration This study was carried out from January 2023 until March 2024.

1.3 Ethical Approval Ethical approval (REC/09/2021(FB/56) dated 17 December 2021 was obtained from the Universiti Teknologi MARA Research Ethics Committee (UiTM REC) to carry out the study at Tourmaline Postgraduate Dental Clinic, Faculty of Dentistry, UiTM. This study was conducted by following the ICH Clinical Practice Guidelines, Malaysia Good Clinical Practice Guidelines and the Declaration of Helsinki. (Appendix 1). Informed consent procedures were detailed, outlining participant recruitment methods and the process by which participants were informed about the study's purpose, risks, benefits, confidentiality measures, and their right to withdraw.

1.4 Reference Population Orthodontic patients requiring fixed appliance treatment involving extractions of at least one premolar in each quadrant with moderate to high anchorage demand.

1.5 Source Population Registered patient attending clinics in Faculty of Dentistry UiTM who require fixed appliance with moderate to high anchorage demand.

1.6 Sample calculation The sample size calculation was done by using G-power analysis (version 3.1.9.7) based on objectives and the findings of the related studies

1.7 Randomisation and allocation Were done in 2 stages, first stage was to allocate the patient into group 1 ( calcium chloride and control) Group 2 ( acid etch and control). Following that, patient were checked for dominant chewers, and to undergo randomisation for allocation of left and right.

Allocation were randomised by block of two for first and second stage.

1.8 Blinding Patient, clinician and statistician were blinded.

1.9 Preparation of OMI OMI will be sterilised first, and immersed in hydrochloric acid at 65°C for 20 minutes, and to be dried in oven. For acid etch, the OMI will be stored in the vacuum sealed vial. For calcium chloride, it will be immersed in 1.0M Calcium Chloride in 4°C storage.

1.10 Clinical 1.4mmx 8mm OMI was inserted between maxillary first molar and second premolar by 2 experienced and callibrated clinician (MMD and MNMS) OMI was inserted 10mm from the bracket slot and tied with metal ligature to maxillary first molar and second premolar as indirect anchorage during treatment. OMI will be removed once the canine is already in class I. Maximum insertion torque is measured by MTT03-50ZU (Mark-10, Copiague,NY.

At day 1,7 and month 3 after insertion, OHIP-14 will be administered via google form to evaluate patient's quality of life. At month 1, 3 and 6, the success of the OMI will be assessed. Success is defined as the ability to maintain the anchorage . Maximum removal torque ( using MTT03-50ZU (Mark-10, Copiague,NY,) is measured after canines are in class I.

1.11 Following removal of the OMI The OMI is assessed under the scanning electron microscop (SEM)

1.12 Statistical analysis Analysis is depending on the distribution of data.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 18 and 40 years
2. Good oral hygiene1
3. Patients prescribed with fixed appliance who require extraction of at least one premolar at each quadrant.
4. Moderate anchorage demand criteria
5. Class II/1 incisor relationship

Exclusion Criteria:

1. History of previous orthodontic treatment
2. Patient who requires combination of orthodontic and orthognathic surgery
3. Medically compromised2 or patients who is taking any medication that interferes with bone metabolism.
4. Presence of craniofacial syndromes or clefts
5. Active periodontal disease
6. Poor oral hygiene prior to orthodontic treatment
7. Smoking3

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Maximum insertion torque and removal torque | During procedure
  Measurement of torque during insertion and removal of the mini implant. The higher the Ncm value, the higher is the stability of the mini implant. The values are directly proportionate to the stability.

SECONDARY OUTCOMES:
Oral Health Quality of Life | During procedure
  OHIP-14 simplified questionaire were distributed to patients to assess the quality of life during treatment with Mini implant. This questionnaire was given at the end of day 1, day 7 and month 3. OHIP-14 is based on summation of score, the higher the score, the worse the quality of life was for the patient. This also assessed the pain score, on VAS scale, the higher the score, the more pain was experienced by patients.
The surface roughness characteristics of the mini implant | at the end of the study at 12 months
  The roughness assessed by Scanning electron microscopy (SEM). The shape and the distribution of bony spicules were assessed. Shapes were assessed if they were of the same shape or sizes. The distributions were assessed in terms of whether it was uniform and homegenous or scattered.
Success rate of mini implant | From enrolment to 6 months
  The success rate within 1 , 3 and 6 months. The success of mini implant is observed by characterised by, no notable mobility and ability to sustain orthodontic force during the treatment. Mobile mini implant that is movable by 3mm are considered as fail mini implant

CONTACTS AND LOCATIONS:
Overall Officials: MARYATI MD DASOR, Study Chair — UNIVERSITY TECHNOLOGY MARA MALAYSIA
Locations (1):
- University Technology Mara Malaysia, Sungai Buloh, Selangor, Malaysia